CLINICAL TRIAL: NCT03556670
Title: Active Workplace Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland State University (Other)
Responsible Party: Principal Investigator, Brad Wipfli, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Active Workplace Study
Record Dates: First submitted 2018-05-03; First posted 2018-06-14 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Sedentary Lifestyle; Occupational Exposure; Health Behavior; Safety Issues
MeSH Terms: conditions — Sedentary Behavior; Health Behavior

STUDY DESIGN:
Intervention Model Description: There are two study conditions: intervention and control. Organizations will be randomized to conditions.
Who Masked: Participant
Masking Description: Participants will be aware that they're part of a study, but will be masked as to whether their worksite is an intervention or control site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Worker Health Intervention (Experimental)
  Interventions: Behavioral: Total Worker Health
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Total Worker Health — The intervention combines organizational and individual level strategies. Participants will be given access to pedal stands, health and safety messaging, and other environmental modifications. Intervention activities that participants could be asked to complete include: computer based training, goal setting and behavioral self-monitoring, scripted team-based health and safety discussions, and team competitions with pedal stands. Supervisor participants could additionally be asked to complete additional computer based training, goal setting and behavioral self-monitoring of supportive behaviors, and inter-supervisor observations. The intervention is six-months in duration.
  Arms: Total Worker Health Intervention
Other: Control — Usual practice control
  Arms: Control

SUMMARY:
Exposure to sedentary work is an occupational hazard with significant health and safety consequences. Sedentary behavior is an independent predictor of heart disease, diabetes, early mortality, and accounts for the majority of the increase in obesity in the US. Prolonged sitting, common in modern sedentary work environments, contributes to increases in musculoskeletal pain, injuries, and detrimental changes in physiological functioning. Call center employees, who are among the most sedentary workers in the US, area priority population for Total Worker Health interventions. This project is designed to substantially improve health, safety, and well-being in call center employees, including physiological outcomes that contribute to chronic diseases.The study tests whether a Total Worker Health oriented intervention is more effective than usual practices for increasing the utilization of health and safety resources and improving worker health and safety. Study results will have implications for over 30 million sedentary workers in the US.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how a Total Worker Health intervention targeting sedentary behavior among call center employees improves the health, safety, and well-being of sedentary workers. Our primary hypothesis is that a multilevel integrated intervention that follows the Total Worker Health approach will have a stronger impact on primary outcomes (sedentary time and light physical activity at work, musculoskeletal pain, time lost due to injury or illness) compared to a control condition that matches typical worksite practices. To test our hypothesis, we will 1) tailor Total Worker Health intervention components to the call center environment, 2) determine the effects of a 6-month intervention, and 3) measure the durability of intervention effects at 12-month follow-up.

The study will use a randomized control trial design with two conditions: a control condition and a Total Worker Health intervention condition that includes organizational and individual intervention components. Study participants will include employees and supervisors from up to eight call centers. The call centers will be randomly assigned to the two conditions prior to the start of the study. During the study, we will conduct a baseline assessment; implement a six-month intervention; conduct a post-intervention assessment; and conduct a follow-up assessment at twelve months. During each assessment period, study participants in both conditions will complete a survey, physical measures, hemoglobin A1c measurement, and seven days of physical activity data collection with accelerometers. Study participants in both conditions could additionally be asked to complete a measurement for endothelial function during each assessment.

The baseline assessment will occur directly after participant enrollment and consent at each worksite. Both conditions will be given access to portable pedal stands. The intervention condition will have additional environmental alterations including hanging signs throughout the work environment that promote health and safety behaviors; and replacing high calorie and high sugar food and drink options in vending machines and break rooms with fresh fruits, vegetables, and other healthier choices.

Participants in the intervention condition will begin intervention activities. Intervention activities that participants could be asked to complete include: computer based training, goal setting and behavioral self-monitoring, scripted team-based health and safety discussions, and team competitions with pedal stands. Supervisor participants could additionally be asked to complete additional computer based training, goal setting and behavioral self-monitoring of supportive behaviors, and inter-supervisor observations. Participants in the control condition will receive no additional support beyond the provision of pedal stands.

Repeated measures will be collected at baseline, six months, and 12 months. Our primary hypotheses are that the intervention condition will produce greater reductions in sedentary behavior, increases in light physical activity, and reductions in musculoskeletal pain and sick day use than the control condition. To test these hypotheses, we will employ an intent-to-treat strategy using generalized estimating equations in order to use all available data to evaluate group differences in the magnitude of change over time in primary outcomes. The effect of interest for each outcome will be the interaction of condition X time. We will statistically control for confounders by measuring a wide range of demographic and psychological variables that could impact study outcomes. We will test for baseline differences between conditions on these variables using one-way ANOVAs (continuous variables) or chi-squares tests (categorical variables). Variables that differ significantly between groups at baseline will be included as covariates in the generalized estimating equation models of intervention effects over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently working in a participating organization

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sedentary behavior | Change from baseline at 6 months and 12 months
  Sedentary behavior at work measured via accelerometry

SECONDARY OUTCOMES:
Height | Baseline, 6-months, and 12-months
  Height
Body weight | Change from baseline at 6 months and 12 months
  Directly measured body weight
Percent body fat | Change from baseline at 6 months and 12 months
  Directly measured percent body fat via bioelectric impedence
Blood pressure | Change from baseline at 6 months and 12 months
  Direct measurement
Resting heart rate | Change from baseline at 6 months and 12 months
  Direct measurement
Hemoglobin A1c | Change from baseline at 6 months and 12 months
  Direct measurement with Siemens DCA Vantage Analyzer
Endothelial functioning | Change from baseline at 6 months and 12 months
  Direct measurement with EndoPat software and hardware
Depression symptoms | Change from baseline at 6 months and 12 months
  CES-D Short Form Scale
Job Stress | Change from baseline at 6 months and 12 months
  Stress in General Scale
Work Family Conflict | Change from baseline at 6 months and 12 months
  Work Family Conflict Scale
General Life Stress | Change from baseline at 6 months and 12 months
  Perceived Stress Scale
Job satisfaction | Change from baseline at 6 months and 12 months
  Michigan Organizational Assessment Questionnaire job satisfaction scale
Global Health | Change from baseline at 6 months and 12 months
  PROMIS Global Health Scale
Support at work | Change from baseline at 6 months and 12 months
  Survey measure of perceived support from supervisors at work
Dietary behaviors | Change from baseline at 6 months and 12 months
  Frequency of high-calorie food and drink consumption
Physical Activity survey | Change from baseline at 6 months and 12 months
  Healthy Physical Activity Scale
Sleep Quality | Change from baseline at 6 months and 12 months
  Pittsburgh Sleep Quality Index
Sleep Distrubance | Change from baseline at 6 months and 12 months
  PROMIS Sleep Disturbance Scale
Sleep Impairment | Change from baseline at 6 months and 12 months
  PROMIS Sleep Impairment Scale
Safety climate | Change from baseline at 6 months and 12 months
  Safety Climate Scale
Musculoskeletal pain | Change from baseline at 6 months and 12 months
  Survey measure of musculoskeletal pain (Nordic Musculoskeletal Symptoms Questionnaire)
Lost work time | Change from baseline at 6 months and 12 months
  Sick days, tardiness, time lost due to injury and illness, and other work absences
Physical activity accelerometer | Change from baseline at 6 months and 12 months
  Physical activity measured via accelerometry
Occupational Sitting | Change from baseline at 6 months and 12 months
  Occupational Sitting and Physical Activity Questionnaire
Job Turnover Intentions | Change from baseline at 6 months and 12 months
  Job Turnover Intentions Scale
Lost Work Time | Change from baseline at 6 months and 12 months
  Days missed at work due to illness and injury

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will not be routinely provided to other researchers outside of the investigator team. However, requests for specific data from national governmental or international science-based organizations seeking to conduct meta-analyses of such data will be honored. We will make aggregated data from the analyses available to qualified researchers through publications and presentations at scientific meetings. We will make all our quantitative de-identified data available to other scientists after the publication of findings linked to our specific aims outlined in the research plan through the Data Repository or directly if not maintained in the Repository.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Wipfli B, Wild S, Hanson GC, Shea SA, Winters-Stone K, Thosar SS. The active workplace study: Protocol for a randomized controlled trial with sedentary workers. Contemp Clin Trials. 2021 Apr;103:106311. doi: 10.1016/j.cct.2021.106311. Epub 2021 Feb 2. PMID 33539991